CLINICAL TRIAL: NCT01169103
Title: Effect of rhGH Administration on Visceral Adiposity and Markers of Cardiovascular Risk in Obese Adolescent Girls: Phase 2
Brief Title: Effect of Recombinant Human Growth Hormone (rhGH) on Abdominal Fat and Cardiovascular Risk in Obese Girls
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Madhusmita Misra, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009P000861
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: Obesity; Adolescent; Insulin resistance; Growth hormone; Visceral fat; Adolescent obesity
MeSH Terms: conditions — Obesity; Insulin Resistance; Pediatric Obesity | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- recombinant human growth hormone (Experimental): Forty subjects will be randomized to receive either recombinant human growth hormone or placebo.
  Interventions: Drug: recombinant human growth hormone (rhGH)
- Placebo (Placebo Comparator): Forty subjects will be randomized to receive either recombinant human growth hormone or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human growth hormone (rhGH) — Initial rhGH dose 0.4mg administered by subcutaneous injection daily. Dose will be increased to 0.6 mg after one week and then increased to 0.8mg after two weeks.
  Arms: recombinant human growth hormone
Drug: Placebo — Placebo will be administered by daily subcutaneous injections. Sham increases will be used.
  Arms: Placebo

SUMMARY:
Teenagers and adults who are overweight or obese have an increase in fat in the abdomen, which increases their risk for diabetes and heart disease. Reducing abdominal fat is important to reduce risk for diabetes and for heart disease. Overweight teenagers also have low levels of growth hormone compared to normal weight teenagers, and teenagers with the lowest growth hormone levels also have the greatest abdominal fat. In children who are unable to make growth hormone for other reasons, giving back growth hormone leads to a decrease in abdominal fat. We are studying whether giving growth hormone in small doses to overweight teenagers can change body composition. We hypothesize that growth hormone will cause abdominal fat to decrease and reduce the risk markers for diabetes and heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls 13-21 years old with bone age ≥ 14 years
* Overweight girls: Body Mass Index (BMI) greater than the 95th percentile for age
* Waist/Hip ratio ≥ 0.85
* Insulin Like Growth Factor -1 (IGF-1) below -0.5 standard deviations (SD) for pubertal stage or age

Exclusion Criteria:

* Pregnancy (positive pregnancy test) prior to enrollment in the study
* Significant weight gain or loss within 3 months of study (more than 5 kg)
* Use of medications that affect GH or cortisol levels (such as estrogen including oral contraceptive pills, oral glucocorticoids)
* Use of medications such as Meridian and Orlistat
* Presence of diabetes mellitus
* Uncontrolled Thyroid disorders
* Chronic renal insufficiency
* Participation in another simultaneous medical investigation or trial
* Active neoplasm or history of cancer
* Prader-Willi syndrome
* History of scoliosis if bone age is <15 years
* Hypersensitivity to rhGH or constituents of the injections

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Slattery M, Bredella MA, Stanley T, Torriani M, Misra M. Effects of recombinant human growth hormone (rhGH) administration on body composition and cardiovascular risk factors in obese adolescent girls. Int J Pediatr Endocrinol. 2014;2014(1):22. doi: 10.1186/1687-9856-2014-22. Epub 2014 Nov 15. PMID 25435886
- [Derived] Slattery MJ, Bredella MA, Thakur H, Torriani M, Misra M. Insulin resistance and impaired mitochondrial function in obese adolescent girls. Metab Syndr Relat Disord. 2014 Feb;12(1):56-61. doi: 10.1089/met.2013.0100. Epub 2013 Nov 19. PMID 24251951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Massachusetts General Hospital between September 2010 and October 2012 through area pediatric and obesity clinics and advertisements.
Pre-assignment Details: Of the 32 subjects who were screened, 22 were eligible & randomized. 5 subjects were ineligible due to Insulin Like Growth Factor levels above the eligibility limit for pubertal stage or age. 2 were excluded due to planned initiation of medications that were on the exclusion criteria list and 3 voluntarily withdrew consent prior to randomization.
Groups:
- Recombinant Human Growth Hormone: Forty subjects will be randomized to receive either recombinant human growth hormone or placebo/no treatment.
  recombinant human growth hormone (rhGH) : Initial rhGH dose 0.4mg administered by subcutaneous injection daily. Dose will be increased to 0.6 mg after one week and then increased to 0.8mg after two weeks.
- Placebo/no Treatment: Forty subjects will be randomized to receive either recombinant human growth hormone or placebo.
  Placebo : Placebo will be administered by daily subcutaneous injections. Sham increases will be used. Due to expiration of placebo medication, placebo subjects who enrolled after 6/2012 were randomized to no treatment.
Period: Overall Study
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Started | 11 | 11
Completed | 5 | 7
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 8 | 17
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (2.6) | 16.9 (2.1) | 16.6 (2.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Visceral and Subcutaneous Abdominal Adipose Tissue Over 6 Months
Description: Visceral adipose tissue (VAT) and subcutaneous abdominal adipose tissue (SAT) were assessed using single slice MR imaging (MRI)
Time Frame: Baseline and 6 months
Population: Due to scheduling difficulties one no treatment subject did not perform the MRI portion of the study at either the baseline or the 6 month visit.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Number analyzed (Participants) | 5 | 6
mm^2
  Change in VAT | 57 (2993) | 799 (3184)
  Change in SAT | -111 (6078) | 3634 (5161)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; We assumed that mean decrease in visceral fat in our population would be 0.85*standard deviation score (SDS). Therefore, 18 subjects in each group would be required in order for us to have an 81.7% chance of detecting a significant difference in the mean 6-month changes in visceral adiposity between the groups at a 5% significance level by rejecting the null hypothesis that there is no difference in change in visceral fat following administration of rhGH or placebo in obese adolescent girls; Test type: Superiority or Other; p = 0.70, t-test, 2 sided
Statistical Analysis 2: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Change in SAT p-value; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

2. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) Score
Description: Homeostasis model assessment of insulin resistance (HOMA-IR) was used as a validated measure of insulin resistance. A 2-hour Oral Glucose Tolerance Test (OGTT) using 1.75 gram/kilogram of oral glucose (maximum 75 gram) will be performed at baseline and six months after administration of rhGH/placebo/ no therapy. Fasting insulin and glucose will be used to determine HOMA-IR: [fasting glucose (mmol/l) x fasting insulin (µU/ml)]/22.5]
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Number analyzed (Participants) | 5 | 7
HOMA-IR score | -0.52 (2.63) | -2.92 (8.23)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Changes in Lipid Panel
Description: Lipid profile will be obtained using established methods. Total Cholesterol, Triglycerides, LDL and HDL measurements will be obtained at baseline, and then at the six-month visits to determine the rate at which lipid measures change with rhGH therapy
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Number analyzed (Participants) | 5 | 7
mg/dL
  Change in Total Cholesterol | -37.8 (23.9) | -8.6 (15.5)
  Change in Triglycerides | -27.8 (46.8) | 6.1 (58.4)
  Change in LDL | -25.8 (12.8) | -10.7 (11.9)
  Change in HDL | -6.6 (6.1) | 1 (5.1)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Change in Total Cholesterol p-value; Test type: Superiority or Other; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Change in Triglyceride p-value; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Change in Low-density lipoprotein p-value; Test type: Superiority or Other; p = 0.062, t-test, 2 sided
Statistical Analysis 4: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Change in High-density lipoprotein p-value; Test type: Superiority or Other; p = 0.0396, t-test, 2 sided

4. Primary Outcome: Change in High-sensitivity C-reactive Protein (Hs-CRP) Over 6 Months
Description: As a marker of cardiovascular risk, hs-CRP will be assessed at baseline and 6 months to assess the rate at which hs-CRP levels change with rhGH therapy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Number analyzed (Participants) | 5 | 7
mg/L | -0.77 (2.4) | -0.09 (1.8)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Test type: Superiority or Other; p = 0.58, t-test, 2 sided

5. Primary Outcome: Change in Soluble Intercellular Adhesion Molecule-1 (sICAM) Over 6 Months
Description: Soluble intercellular adhesion molecule-1 (sICAM) was used as a surrogate marker of cardiovascular risk
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Number analyzed (Participants) | 5 | 7
ng/mL | -22.2 (30.3) | 21.1 (33.3)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo/no Treatment; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Recombinant Human Growth Hormone | Placebo/no Treatment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 10/11 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Human Growth Hormone (N=11) | Placebo/no Treatment (N=11)
Impaired Glucose Tolerance (Endocrine disorders) | 2 | 4 — Impaired Glucose Tolerance (IGT) on 75 Gram 2 Hour Oral Glucose Tolerance Test (OGTT). IGT determined by fasting glucose level > 100 mg/dL or > 140 mg/dL at 2 hours post glucose load
Polyuria/Polydipsia (Endocrine disorders) | 1 | 3
HbA1c > 6.4% (Endocrine disorders) | 1 | 0
Headache (General disorders) | 4 | 3
Nausea with vomiting (Gastrointestinal disorders) | 1 | 0
Nausea without vomiting (Gastrointestinal disorders) | 3 | 0
Dizziness without Headace (General disorders) | 0 | 1
Blurry Vision (Eye disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Change in Menstrual Flow (Endocrine disorders) | 3 | 2
Fatigue (Endocrine disorders) | 0 | 2
Bruising/Irritation at Injection Site (Injury, poisoning and procedural complications) | 2 | 2
Bruising/Irritation at Blood Sampling Site (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
ED visit for wheezing with URI (General disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Nasal Congestion (Infections and infestations) | 1 | 0
Eczema (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No